CLINICAL TRIAL: NCT01388998
Title: External Pressure Applied on the Caval Vein and Its Effects on Difference in Pulse Pressure (dPP) and Pleth Variability Index (PVI)
Brief Title: Fluid Management Study to Evaluate Changes in Intravascular Volume After Applying Various Pressure Levels on the Caval Vein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Lydia T. Strys, M.D., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 837.308.10(7317)
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Intravascular Volume; Respiratory Changes
Keywords: fluid management; fluid therapy; dPP; difference in pulse pressure; PVI; pleth variability index; external pressure applied on the caval vein
MeSH Terms: interventions — Blood Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Changes of difference in pulse pressure and plethysmography after applying various pressure levels on the caval vein — Following hepatic resection, a fitting area for pressure application on the caval vein will be identified by the attending surgeon. Baseline assessments of hemodynamic and heart-lung interaction parameters will be taken. Thereafter the surgeon will apply three different pressure levels (2 N, 5 N, 10 N) at random with a force gauge (Fa. ATP Messtechnik, Ettenheim, Germany). Assessment of the parameters will be performed after 2 minutes of pressure application by an investigator, unaware of the pressure applied. After each pressure application 5 minutes will be waited to assure hemodynamic recovery.

SUMMARY:
Fluid therapy optimization in the perioperative period has been considered as major contributor to improve oxygen delivery. A recent, noninvasive approach to estimate fluid requirements in the anesthetized patient with arterial line is the assessment of difference in pulse pressure (dPP). Intraoperative fluid management by dPP is a goal-directed fluid management approach to avoid both hypervolemia and hypovolemia. However, several clinical factors may impede dPP measurements. Surgical manipulations in abdominal procedures may interfere with hemodynamic stability due to obstruction of the caval vein. Physiological considerations make us hypothesize that only intense pressure impedes caval blood flow and thus hemodynamics and dPP. Therefore, the investigators want to assess those changes after standardized application of three different pressure levels (2 N, 5 N, 10 N) on the caval vein.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective hepatic surgery procedures (hemihepatectomy) qualifying for arterial line

Exclusion Criteria:

* pregnancy
* cardiac insufficiency (NYHA 4, EF < 25 %)
* coronary (CCS 4)
* coagulopathy
* symptoms of infection or sepsis
* malignant hyperthermia
* porphyria
* oesophageal varicose veins
* absence of sinus rhythm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change of dPP from start of intervention to 2 minutes after start of the intervention | Application of pressure for 2 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lydia T. Strys, MD, Principal Investigator — Universitaetsmedizin - Johannes Gutenberg University Mainz (Department of Anesthesiology); Dorothea Closhen, MD, PhD, Principal Investigator — Universitaetsmedizin - Johannes Gutenberg University Mainz (Department of Anesthesiology); Gunther Pestel, MD, PhD, Study Director — Universitaetsmedizin - Johannes Gutenberg University Mainz (Department of Anesthesiology)
Locations (1):
- Universitaetsmedizin - Johannes Gutenberg University Mainz (Department of Anesthesiology), Mainz, Germany